CLINICAL TRIAL: NCT02906852
Title: Prospective Observational Study to Evaluate the Performance of Inivata Liquid Biopsy Analysis Compared With Standard Tissue Biopsy Analysis for Detection of Genomic Alterations in Patients With Advanced Non-small Cell Lung Cancer.
Brief Title: Concordance of Inivata Liquid Biopsy With Standard of Care Tissue Testing
Status: Completed | Type: Observational
Sponsor: Inivata (Industry)
Collaborators: Vector Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: INI001
Record Dates: First submitted 2016-09-02; First posted 2016-09-20 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A 40ml blood sample will be taken, from which Plasma and ultimately DNA will be prepared.
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate the performance of Inivata liquid biopsy analysis compared with standard tissue biopsy analysis for detection of genomic alterations in patients with advanced lung cancer.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the performance of Inivata liquid biopsy analysis compared with standard tissue biopsy analysis for detection of genomic alterations in patients with advanced lung cancer. Once selected for the study and with full informed consent, patients will have a blood draw to allow the detection of cancer-related genomic alterations that are detectable within the blood sample. These results will be compared to results obtained from genomic profiling via standard tissue biopsy taken as part of routine care to help determine whether such 'liquid biopsies' can be used to guide treatments in future patients. The results of the liquid biopsy will not be used to guide treatment decisions in study participants.

In addition there is data-collection of treatments received for non small cell lung cancer and the response to these treatments during the first 6 months post tissue and blood analysis, though no additional visits or procedures are required for the patient beyond the initial blood draw.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed and dated informed consent to participate in the study must be given by the patient in accordance with 21 CFR Part 312, the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6, and applicable regulations, before completing any study-related procedures.
* Male and female patients aged 18 years and over diagnosed with stage IIIb/IV non-squamous NSCLC.
* Arms A and B: Patients intended to initiate first-line treatment according to standard guidelines. Note, a patient is eligible to receive sterotactic radiosurgery (no whole-brain radiotherapy). Arm C: Patients who are at a second-line treatment setting or greater may participate. Note, a patient may be included if they have metastatic brain lesions. Arms A, B, C: If enrolled in a treatment clinical trial, patients may also enroll in this study if all eligibility criteria are met.
* Arm A only: Patients intended to initiate first-line treatment according to standard guidelines who plan to have or have had a recent tumor tissue biopsy taken for molecular profiling as part of their standard of care.
* Patient must understand and be able, willing and likely to fully comply with all study procedures and restrictions.

Exclusion Criteria:

* Patients who have received any approved or experimental cancer therapy since their most recent NSCLC tissue biopsy (Arms A and B)
* Patients who have any other prior metastatic or current second primary cancer (Arms A and B)
* Patient who has a severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients aged 18 years and over diagnosed with stage IIIb/IV non-squamous NSCLC, who are intended to initiate first-line treatment according to standard guidelines, or having recently progressed on first-line EGFR or ALK directed therapy and being considered for further therapy.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Concordance in the detection of molecular abnormalities using Inivata's liquid biopsy panel with detection using standard of care tissue biopsy analysis | 1 year

SECONDARY OUTCOMES:
Detection: sensitivity and specificity of molecular abnormalities using Inivata liquid biopsy panel relative to standard of care tissue biopsy analysis | 1 year
Proportion of NSCLC patients eligible for targeted therapy based on liquid biopsy analysis as an evaluation of feasibility molecular stratification, compared to standard of care alone | 1 year
Progression free survival (PFS) rate over 6 months | 1 year
Overall survival (OS) rate over 6 months | 1 year

OTHER OUTCOMES:
Relationship of clinical response to therapy with mutation allele frequency (MAF) cutoff in Inivata liquid biopsy assay | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, MD, Principal Investigator — Washington University School of Medicine; Edward Kim, MD, Principal Investigator — Atrium Health Levine Cancer Institute; Clive Morris, MD, Study Director — Inivata
Locations (35):
- United States (35):
  - Facey Medical Foundation, Mission Hills, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Eastern CT Hematology Oncology, Norwich, Connecticut
  - Christiana Care Health Services Inc, Newark, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mid-Florida Hematology and Oncology Centers, Orange City, Florida
  - Swedish Covenant Hospital, Chicago, Illinois
  - Edward M Kaplan, MD & Associates, Skokie, Illinois
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Norton Healthcare Inc, Louisville, Kentucky
  - Christus Cancer Treatment Center, Shreveport, Louisiana
  - Berkshire Hematology Oncology Services, Pittsfield, Massachusetts
  - Henry Ford Allegiance Health, Jackson, Michigan
  - Park Nicolett, Saint Louis Park, Minnesota
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - Boone Hospital Center, Columbia, Missouri
  - Washington University (St. Louis), St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Northshore Hematology Oncology, East Setauket, New York
  - Northern Westchester Hospital Association, Mount Kisco, New York
  - East Carolina University, Greenville, North Carolina
  - Levine Cancer Center, Mint Hill, North Carolina
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - Trinity Cancer Center, Minot, North Dakota
  - Providence Health and Services, Portland, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Carolina Blood and Cancer Care, Rock Hill, South Carolina
  - The West Clinic, Germantown, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Thomas Spann Clinic Oncology, Corpus Christi, Texas
  - Hope Cancer Center of East Texas (Tyler Hem Onc), Tyler, Texas
  - Virginia Cancer Institute, Richmond, Virginia
  - Providence Regional Medical Center, Everett, Washington
  - University of Washington (Swedish General), Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No